CLINICAL TRIAL: NCT01817478
Title: The Influence of Hospital Environment on Eyes Infections in Medical Staff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0093-12-ZIV
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Eye Infections
Keywords: conjunctival flora
MeSH Terms: conditions — Eye Infections

ARMS (1):
- medical staff (Experimental)
  Interventions: Other: microbiologic sample

INTERVENTIONS:
Other: microbiologic sample

SUMMARY:
The investigators want to find out if there is any difference between the microbiotic flora lining the conjunctiva of medical staff that work in the hospital and others who do not work in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* healthy medical workers.

Exclusion Criteria:

* any ocular disease.
* previous ocular surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
significant difference in the bacterial flora of conjunctiva | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel